CLINICAL TRIAL: NCT05480930
Title: Novel Approach to Improve Patient Care and Diarrheal Disease Research Using Mobile Technology in Haiti
Brief Title: Improving Nighttime Access to Care and Treatment; Part 4-Haiti
Acronym: INACT4-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB202201220; R21TW012332 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-07-29 (Actual); Last update posted 2025-06-30 (Actual); Status verified 2025-06

CONDITIONS: Telemedicine; Pediatrics
Keywords: digital clinical decision support
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: This study is an interrupted time series trial where the pre-intervention period will employ existing paper clinical decision support tools and the intervention period will employ a new digital clinical decision support tool. A small fraction of participants will participate in both the pre-intervention and post-intervention periods but most will only participate in one.
Who Masked: Participant
Masking Description: Participants who are consulted/examined by telephone only will be masked to which arm they are participating in. Participants who are consulted/examined in-person will not be explicitly informed of the study arm but will be able to observe if the provider is using paper forms or an electronic device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paper-based clinical decision support tool (Active Comparator): Providers at the TMDS will use the existing paper-based clinical decision support tools to consult/examine patients.
  Interventions: Other: paper-based clinical decision support (dCDS) tool
- digital clinical decision support (dCDS) tool (Experimental): Providers at the TMDS will use the new digital clinical decision support (dCDS) tool to consult/examine patients.
  Interventions: Other: digital clinical decision support (dCDS) tool

INTERVENTIONS:
Other: paper-based clinical decision support (dCDS) tool — The paper based clinical decision support tools currently employed at the TMDS that are used to triage, assess and generate treatment plans for pediatric patients.
  Arms: paper-based clinical decision support tool
Other: digital clinical decision support (dCDS) tool — The intervention is a digitized version of the paper based clinical decision support tools currently employed at the TMDS that are used to triage, assess and generate treatment plans for pediatric patients.
  Arms: digital clinical decision support (dCDS) tool

SUMMARY:
Children in resource-limited settings who develop illness at night are often isolated from care, resulting in progression to an emergency. A telemedicine and medication delivery service (TMDS) is a viable healthcare delivery option to bridge the gap in nighttime care. This interrupted time series study (pre/post) will evaluate a digital clinical decision-support (dCDS) tool. The objective is to assess if the tool is associated with an improvement in guideline adherence by TMDS providers.

DETAILED DESCRIPTION:
Acute respiratory infection and diarrheal disease are the two leading causes of pediatric death between 1 month and 5 years of age globally. These common problems have well-established low-cost treatments. However, these treatments are most effective when administered early which is difficult in resource-limited settings, especially at night. Based on five years of formative NIH-funded research, the team has built a Telemedicine and Medication Delivery Service (TMDS) in Haiti to improve nighttime access to care and treatment for children called MotoMeds. The strategic plan is to design, deploy and evaluate MotoMeds by conducting four clinical studies titled Improving Nighttime Access to Care and Treatment (INACT1/2/3/4) in Haiti. INACT1-H was a needs assessment (2018-2019), INACT2-H was a pre-pilot deployment of MotoMeds that compared the congruence of clinical assessments at the call-center to in-person household assessments by providers (2019-2020), and INACT3-H was a pilot of a scalable model of MotoMeds that had provider assessment only at the call-center for most non-severe cases and had provider assessment at both the call-center and household for some non-severe/ moderate cases. In addition, the central call center serviced a geographically distant delivery zone, demonstrating proof of concept for a fully scaled model. INACT4-H will evaluate a digital clinical decision support (dCDS) tool designed for use at a pediatric TMDS in an interrupted time series study. The pre-intervention is use of the existing paper CDS tool and the intervention is use of the dCDS tool. This initiative is significant because it uses telemedicine and medication delivery to address one of the most fundamental challenges in pediatrics early access to pediatric healthcare.

ELIGIBILITY:
Inclusion criteria for child, parent/guardian participants:

* Children 10 years of age or younger with an acute illness
* Parent/guardian contacts the TMDS in regards to the illness during hours of operation
* Parental/guardian agreement to a waiver of documentation of consent when contact is by phone only OR written consent/assent at the household from the parent/guardian and child (7yrs and older) for participants who receive a household visit.

Exclusion criteria for child, parent/guardian participants:

* No consent

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7124 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in provider guideline adherence rates at the call center between use of the paper and digital clinical decision support tools (CDS). | Two 16 month intervention periods less the 2 week wash out.
  We will evaluate the change in rates of provider guideline adherence at the call center between the 16 month period (minus 2 week wash out) where the existing paper CDS tools are used and the 16 month period (minus 2 week wash out) where the new digital CDS tools are used. Guideline adherence will be measured using the following features of the assessment and plan; severity determination and danger signs, provider household visit determination, and antibiotic and zinc prescriptions.

SECONDARY OUTCOMES:
Enumeration of clinical status of participants at 10-day follow up | 10 days
  All families will receive a follow-up call at 10 days post initial call to MotoMeds. The family will be asked about the clinical status of the child with regards to the initial medical complaint (resolved, better, same, worse, died).
Change in call duration between use of the paper and digital clinical decision support tools (CDS). | From time incoming call is answered until treatment plan has been explained (approximately 10 to 20 minutes).
  Call duration is defined as the time elapsed from once the provider starts consulting the patient (filling out the case report form or face sheet) until the provider finishes the assessment and has communicated the treatment plan to the caller (prior to the consent process). The mean call duration while using the paper CDS will be compared to the mean call duration while using the digital CDS tool.
Change in time to medication delivery between use of the paper and digital clinical decision support tools (CDS). | From time incoming call is answered until medication is delivered to the participant's home (approximately 45-120 minutes).
  Time to medication delivery is defined as the time from once the provider starts consulting the patient (filling out the case report form or face sheet) until the driver (or driver and provider) arrives at the patient's home for delivery. The mean time to delivery while using the paper CDS will be compared to the mean time to delivery while using the digital CDS tool.

OTHER OUTCOMES:
Change in provider guideline adherence rates at the household between use of the paper and digital clinical decision support tools (CDS). | Two 16 month intervention periods less the 2 week wash out.
  We will evaluate the change in rates of provider guideline adherence at the household between the 16 month period (minus 2 week wash out) where the existing paper CDS tools are used and the 16 month period (minus 2 week wash out) where the new digital CDS tools are used. Guideline adherence will be measured using the following features of the assessment and plan; severity determination and danger signs, provider household visit determination, and antibiotic and zinc prescriptions.
Qualitative feedback from TMDS providers | Approximately 1 hour
  Qualitative feedback from the provider perspective framed with respect to content, usability of the user-interface (e.g., haptic vs typed data entry, navigation), satisfaction and technical challenges (connectivity, malfunctions, inter-operability).

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Nelson, MD PhD, Principal Investigator — University of Florida
Locations (1):
- CV Foundation, Gressier, Ouest, Haiti

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share a de-identified data set in a data depository such as Dryad.
Supporting Information: Study Protocol
Time Frame: The data will likely be made available within 1 year of the conclusion of the study.
Access Criteria: The de-identified dataset will be deposited in a publicly available data depository such as Dryad.

REFERENCES:
- See also: MotoMeds TMDS website at the University of Florida — https://nelson.research.pediatrics.med.ufl.edu/motomeds/